CLINICAL TRIAL: NCT01427413
Title: Identification and Standardization of a Method That Would Allow the Study of the Metabolic Profile of Blastocoele Lays the Foundation to Assess Blastocyst Metabolomic Profile and Its Relation With Embryo Morphology and Embryo Implantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cervesi Hospital, Cattolica, Italy (Other)
Collaborators: Università degli Studi La Tuscia (Unknown); Tecnobios Riproduzione (Unknown); Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Palini Simone, Embryologist, Cervesi Hospital, Cattolica, Italy
Other Study IDs: SS4e
Record Dates: First submitted 2011-08-29; First posted 2011-09-01 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2020-07

CONDITIONS: Blastocoele Fluid
Keywords: blastocoele fluid; mass spectrometry; metabolomics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blastocoele fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hyper1: Only patients who achieved hyperstimulation pathology after external administration of gonadotrophin during IVF treatment

SUMMARY:
While the number of assisted reproduction cycles increases worldwide, the introduction of actual technological improvements in the ability to quickly and non-invasively identify the best embryos for transfer still represents a critical goal for reproductive medicine. Indeed, embryo assessment is currently performed through the analysis of morphology and cleavage rate. Recent studies have sought to identify a correlation between qualitative-quantitative profiles of small molecules of metabolic interest and the outcome of embryo transfer. Some of these molecules seem to be best suited for this purpose, including glucose, lactate, pyruvate or amino acid levels. Approaches relying on both optical and non-optical spectroscopy have been proposed to non-invasively monitor the embryo culture media. However, the non-invasive approach only offers an indirect strategy to monitor embryos and a turn-around solution to bypass the limits of detection of these analytical techniques. In this paper the investigators pave the way for direct assessment of embryos through the mass spectrometry-based analysis of blastocoele fluid, which is withdrawn from the blastocoele cavity prior to cryostorage of blastocysts. The investigators show how it is possible to detect most of the already documented metabolites of interest right at the very heart of the blastocyst, without disrupting the workflow of a classic laboratory pipeline.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian hyperstimulation disease
* Blastocyst formation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the patients that are unable to be subjected to embryo transfer due to her ovarian hyperstimulation. In those cases the embryos will be vitrified and during this procedure we collapse the blastocyst sucking the fluid.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2022-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
standardize the method of aspiration | 2 months
  The method for blastocyst micropuncturing and aspiration of blastocoel fluid is according also to the last literature about blastocyst vitrification. In brief, expanded day 5 blastocysts were removed from culture and transferred to a 30 nl droplet of pre-warmed Hepes buffer.
  An injection pipette was introduced avoiding contaminations through the trophectoderm, and blastocoel fluid was aspirated until the blastocyst had fully collapsed around the pipette. The retrieved fluids were expelled into new purified water drops and frozen at -80°C alongside 0.5 nl control droplets of purified water.
metabolite detection | 6 months
  metabolite detection through rapid resolution reversed phase (RR-RP) high performance liquid chromatography (HPLC)-mass spectrometry (MS). From sample volumes as low as 0.5 nl we could detect and quantify against external standards a group of metabolites, whose roles in blastocyst development and embryo metabolism have long been postulated. The list included i) ATP adenosine triphosphate ; ii) glucose-6-phosphate; iii) lactate; iv) NAD+ nicotinamide-adenine dinucleotide+ and v) NADH and vi) NADPH nicotinamide-adenine dinucleotide phosphate; vii) 6-phosphogluconic acid; viii) glutamic acid and ix) α-ketoglutarate.

SECONDARY OUTCOMES:
analysis of the correlation between blastocyst morphology and metabolic profile in the blastocoele fluid | 1 year
  blastocyst classify according to morphological criteria in the book "Atlas of Human Blastocyst" by L. Veeck and associate, to each morphological class a characteristic metabolic profile, in order to scientifically validate the observational and objective criteria up to now used in our lab

CONTACTS AND LOCATIONS:
Overall Officials: Simone Palini, biology, Study Director — Cervesi Hospital, Cattolica, Italy
Locations (1):
- Cervesi Hospital, Cattolica, Rimini, Italy